CLINICAL TRIAL: NCT03728933
Title: A Remote, Double-Blind, Randomized, Placebo-Controlled Study of Rotigotine Transdermal System in Adolescent Subjects With Idiopathic Restless Legs Syndrome
Brief Title: A Study of Rotigotine Patch in Adolescent Subjects With Restless Legs Syndrome of Unknown Cause
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision; Not a safety decision
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP1006
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-09

CONDITIONS: Restless Legs Syndrome
Keywords: RLS; Rotigotine; Neupro
MeSH Terms: conditions — Restless Legs Syndrome | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 2 milligram/24 hours rotigotine (Experimental): Subjects randomized to this arm will be initiated on 1 milligram (mg)/24 hours (h) rotigotine and up-titrated to a maximum of 2 mg/24 h rotigotine, which is the assigned dose level throughout the 12-week Maintenance Period.
  Interventions: Drug: Rotigotine 1 milligram/24 hours; Drug: Rotigotine 2 milligram/24 hours
- 3 milligram/24 hours rotigotine (Experimental): Subjects randomized to this arm will be initiated on 1 milligram (mg)/24 hours (h) rotigotine and up-titrated to a maximum of 3 mg/24 h rotigotine (1 mg/24 h patch + 2 mg/24 patch at the same time), which is the assigned dose level throughout the 12-week Maintenance Period.
  Interventions: Drug: Rotigotine 1 milligram/24 hours; Drug: Rotigotine 2 milligram/24 hours
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive matching placebo patches to maintain the blinding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rotigotine 1 milligram/24 hours — Pharmaceutical Form: transdermal patch Route of administration: transdermal use Concentration: Application of rotigotine transdermal patch with 1 milligram (mg)/24 hours (h) (5 square centimeter (cm^2) patch size).
  Other Names: Neupro
  Arms: 2 milligram/24 hours rotigotine; 3 milligram/24 hours rotigotine
Drug: Rotigotine 2 milligram/24 hours — Pharmaceutical Form: transdermal patch Route of administration: transdermal use Concentration: Application of rotigotine transdermal patch with 2 milligram (mg)/24 hours (h) (10 square centimeter (cm^2) patch size).
  Other Names: Neupro
  Arms: 2 milligram/24 hours rotigotine; 3 milligram/24 hours rotigotine
Drug: Placebo — Pharmaceutical Form: transdermal patch Route of administration: transdermal use Concentration: not applicable
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy of rotigotine against placebo in adolescent subjects with idiopathic Restless Legs Syndrome (RLS) over a 12-week maintenance period and to investigate the safety and tolerability of rotigotine in adolescent subjects with idiopathic RLS.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, and is >=13 and <18 years of age at Baseline
* Subject's Restless Legs Syndrome (RLS) symptoms cause significant daytime symptoms or significant distress or impairment in social, occupational, educational, or other important areas of functioning by the impact on sleep, energy/vitality, daily activities, behavior, cognition or mood
* At Baseline, subject has a score of >=15 on the International Restless Legs Rating Scale (IRLS) (indicating moderate-to-severe RLS)
* At Baseline, subject scores >=4 points on the Clinical Global Impressions (CGI) Item 1 assessment (indicating at least moderately ill)
* Subjects who are receiving supplemental iron have been on a stable dose for at least 1 month prior to Screening
* Female subjects must be surgically incapable of childbearing, or effectively practicing an acceptable method of contraception (oral/parenteral/implantable hormonal contraceptives, intrauterine device, or barrier and spermicide). Abstinence is an acceptable method. Subjects must agree to use adequate contraception during the study and for 4 weeks after their final dose of study medication.

Exclusion Criteria:

* Subject has a serum ferritin level below the lower limit of normal at Visit 1/Screening
* Subject has a hemoglobin level below the lower limit of normal at Visit 1/Screening
* Subject has had previous treatment with dopamine agonists or L-dopa within 7 days prior to Visit 2/Baseline
* Subject has any medical or psychiatric condition, which in the opinion of the investigator, would jeopardize or compromise the subject's well-being or ability to participate in this study
* Subject is pregnant or nursing
* Subject is not willing to abstain from caffeine after 4 pm each evening within 7 days prior to Visit 2/Baseline and for the duration of the study
* At Visit 1/Screening, subject has symptomatic orthostatic hypotension with a decrease of blood pressure (BP) from supine to standing position of >=20 mmHg in systolic blood pressure (SBP) or of >=10 mmHg in diastolic
* Subject has secondary Restless Legs Syndrome (RLS) (eg, due to renal insufficiency [uremia], iron deficiency, or rheumatoid arthritis)
* Subject has a lifetime history of suicide attempts (including actual attempt, interrupted attempt, or aborted attempt), or had suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening (Visit 1)
* Subject is taking a prohibited concomitant medication. Prohibited concomitant medication must have been discontinued at least 2 weeks prior to Screening (Visit 1)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (1):
- Sp1006 101, Culver City, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in December 2018 and concluded prematurely in July 2022.
Pre-assignment Details: The Participant Flow refers to the Randomized Set.
Groups:
- Placebo: Participants randomized to this arm received placebo as a comparator matched to rotigotine during 3 week titration period and is continued throughout the 12-week Maintenance Period.
- Rotigotine 2 mg/24h: Participants randomized to this arm were initiated on 1 milligram (mg)/24 hours (h) rotigotine and up-titrated to a maximum of 2 mg/24 h rotigotine during 3 week titration period and the same dose is continued throughout the 12-week Maintenance Period.
- Rotigotine 3 mg/24h: Participants randomized to this arm were initiated on 1 mg/24 h rotigotine and up-titrated to a maximum of 3 mg/24 h rotigotine during 3 week titration period and the same dose is continued throughout the 12-week Maintenance Period.
Period: Overall Study
Arm/Group | Placebo | Rotigotine 2 mg/24h | Rotigotine 3 mg/24h
Started | 8 | 8 | 7
Completed | 5 | 7 | 6
Not Completed | 3 | 1 | 1
Not completed — Withdrawal by Parent/Guardian | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Randomized Set consisted of all participants from the Enrolled Set who have been randomized.
Groups:
- Rotigotine 2 mg/24h: Participants randomized to this arm were initiated on 1 mg/24 h rotigotine and up-titrated to a maximum of 2 mg/24 h rotigotine during 3 week titration period and the same dose is continued throughout the 12-week Maintenance Period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Rotigotine 2 mg/24h | Rotigotine 3 mg/24h | Total
Number analyzed (Participants) | 8 | 8 | 7 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (1.3) | 16.1 (1.1) | 15.6 (1.0) | 15.7 (1.1)
Age, Customized [Count of Participants; unit: Participants]
  Adolescents (12-17 years) | 8 | 8 | 7 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 2 | 14
  Male | 2 | 2 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 0 | 1 | 0 | 1
  Black | 0 | 0 | 1 | 1
  White | 7 | 7 | 6 | 20
  Other/Mixed | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 8 | 8 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the End of the Maintenance Period in International Restless Legs Rating Scale (IRLS) Sum Score
Description: The IRLS consisted of 10 questions, each scored using a 5-point scale ranging from 0=not present to 4=very severe. The IRLS sum score was calculated by summing up the single scores of all applicable questions, i.e., the total sum score ranged from 0 (no RLS symptoms present) to 40 (maximum severity in all symptoms). A score between 31 and 40, indicates very severe RLS. A score between 21 and 30 indicates severe RLS. A score between 11 and 20 indicates moderate RLS. A score between 1 and 10 indicates mild RLS and a score of 0 means no RLS. A negative change from Baseline indicates improvement.
Time Frame: From Baseline to the end of the Maintenance Period (Day 106)
Population: The Full Analysis Set (FAS) consisted of all participants from the Safety Set who had a valid IRLS score and a valid clinical global impressions (CGI) Item 1 score at Baseline and a valid post-Baseline IRLS score and a valid post-Baseline CGI Item 1 score. Here, Number of Participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rotigotine 2 mg/24h | Rotigotine 3 mg/24h
Number analyzed (Participants) | 5 | 7 | 5
score on a scale | -8.2 (6.8) [lower limit 6.8] | -14.0 (8.2) [lower limit 8.2] | -6.4 (5.8) [lower limit 5.8]

2. Primary Outcome: Change From Baseline in Clinical Global Impressions (CGI) Item 1 to the End of the Maintenance Period
Description: The Clinical Global Impressions Item 1 (Severity of Illness) score ranges from 0 to 7 as follows: 0=not assessed, 1=normal, not ill at all, 2=borderline ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, 7=among the most extremely ill. The CGI Item 1 was completed during an interview between the participant and the investigator or designee. A negative change from Baseline indicates improvement.
Time Frame: From Baseline to the end of the Maintenance Period (Day 106)
Population: The FAS consisted of all participants from the Safety Set who had a valid IRLS score and a valid CGI Item 1 score at Baseline and a valid post-Baseline IRLS score and a valid post-Baseline CGI Item 1 score. Here, Number of Participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rotigotine 2 mg/24h | Rotigotine 3 mg/24h
Number analyzed (Participants) | 5 | 7 | 5
score on a scale | -1.0 (1.4) [lower limit 1.4] | -1.7 (1.1) [lower limit 1.1] | -0.8 (0.8) [lower limit 0.8]

3. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as events that started during the Treatment Period or within 30 days following the end of the Treatment Period (i.e., on or after the date of first patch application and within 30 days following the date of last patch removal + 1 day), or those events where the intensity worsened within this time frame.
Time Frame: From Baseline to Safety Follow-Up (up to Week 20)
Population: The Safety Set consisted of all participants from the Randomized Set (RS) who had at least one patch (rotigotine or placebo) applied.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Rotigotine 2 mg/24h | Rotigotine 3 mg/24h
Number analyzed (Participants) | 8 | 8 | 7
percentage of participants | 87.5 | 87.5 | 71.4

4. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) Leading to Withdrawals
Description: as for outcome 3
Time Frame: From Baseline to Safety Follow-Up (up to Week 20)
Population: The Safety Set consisted of all participants from the RS who had at least one patch (rotigotine or placebo) applied.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Rotigotine 2 mg/24h | Rotigotine 3 mg/24h
Number analyzed (Participants) | 8 | 8 | 7
percentage of participants | 12.5 | 0 | 0

5. Secondary Outcome: Change From Baseline in Restless Legs-6 Rating Scales (RLS-6) to the End of the Maintenance Period
Description: The RLS-6 Rating Scales was designed to assess the severity of RLS and consisted of 6 subscales. The subscales assessed severity of symptoms at the following times of the day/evening: falling asleep, during the night, during the day at rest, and during the day when engaged in daytime activities. In addition, the subscales assessed satisfaction with sleep and severity of daytime tiredness/sleepiness. Scores for each of the 6 subscales ranged from 0 (completely satisfied) to 10 (completely dissatisfied). The change from baseline was derived for each of the subscales and reported in this outcome measure. A negative change from Baseline indicates improvement.
Time Frame: From Baseline to the end of the Maintenance Period (Day 106)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rotigotine 2 mg/24h | Rotigotine 3 mg/24h
Number analyzed (Participants) | 5 | 7 | 5
score on a scale
  Satisfaction with sleep | -1.8 (4.1) [lower limit 4.1] | -4.7 (2.3) [lower limit 2.3] | -2.0 (2.8) [lower limit 2.8]
  Severity: RLS symptoms at falling asleep | -2.8 (3.6) [lower limit 3.6] | -5.6 (1.6) [lower limit 1.6] | -2.8 (1.8) [lower limit 1.8]
  Severity: RLS symptoms during the night | -1.0 (2.5) [lower limit 2.5] | -2.9 (3.0) [lower limit 3.0] | -2.4 (2.2) [lower limit 2.2]
  Severity: RLS symptoms during the day - at rest | -1.4 (1.3) [lower limit 1.3] | -3.6 (3.5) [lower limit 3.5] | -2.4 (2.6) [lower limit 2.6]
  Severity: RLS symptoms during the day-not at rest | -3.8 (1.9) [lower limit 1.9] | -4.3 (3.5) [lower limit 3.5] | -0.4 (1.1) [lower limit 1.1]
  How tired or sleepy during the day | -3.0 (2.8) [lower limit 2.8] | -5.6 (2.1) [lower limit 2.1] | -3.0 (1.9) [lower limit 1.9]

ADVERSE EVENTS:
Time Frame: From Baseline to Safety Follow-Up (up to Week 20)
Description: TEAEs were defined as events that started during Treatment Period or within 30 days following the end of Treatment Period (i.e., on or after the date of first patch application and within 30 days following the date of last patch removal + 1 day), or those events where intensity worsened within this time frame. TEAEs were analyzed for Safety Set.
Arm/Group | Placebo | Rotigotine 2 mg/24h | Rotigotine 3 mg/24h
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 1/7
Other Adverse Events (participants affected / at risk) | 7/8 | 7/8 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | Rotigotine 2 mg/24h (N=8) | Rotigotine 3 mg/24h (N=7)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | Rotigotine 2 mg/24h (N=8) | Rotigotine 3 mg/24h (N=7)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Application site erythema (General disorders) | 1 (2) | 4 (5) | 1 (1)
Application site pruritus (General disorders) | 0 (0) | 3 (3) | 1 (1)
Application site irritation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (2) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Serum ferritin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Thyroid function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transferrin saturation decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (4)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT03728933/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT03728933/SAP_001.pdf